CLINICAL TRIAL: NCT02927639
Title: MyDiaText: Texting the Way to Better Diabetes Control
Brief Title: MyDiaText Text Messaging Intervention for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-013222; T32DK063688-13S1 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive the intervention for 6 months. The intervention will consist of daily text messages sent to the subject's personal mobile device in addition to the usual standard care. Subjects will be incentivized to respond to text messages via a financial reward lottery system. Previously developed text messages based on the ADA behavior goals will be used for this intervention.
  Interventions: Other: MyDiaText
- Control (No Intervention): This group will receive the usual standard of care for 6 months.

INTERVENTIONS:
Other: MyDiaText — The intervention will consist of daily text messages sent to the subject's personal mobile device.
  Arms: Intervention

SUMMARY:
To test a text messaging intervention using MyDiaText and financial incentives to determine whether such an intervention will improve self-reported self-care behaviors in children 12 to 18 years old. The intervention will consist of daily text messages sent to the subject's personal mobile device. Subjects will be incentivized to respond to text messages via a lottery financial incentive. Previously developed text messages based on the American Diabetes Association (ADA) behavior goals will be used for this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes for more than 1 year
* HbA1c greater than or equal to 8% but less than 14%.
* Have been seen in diabetes clinic in the last 6 months
* Owns a personal mobile device with unlimited text messaging plan

Exclusion Criteria:

* Non-English speaking
* Significant cognitive disability or major organ illness
* Hemolytic anemia

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Lipman, PhD, Principal Investigator — CHOP
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 83 | 82 (1 subj was inadvertently enrolled in another interventional study just before enrolling so removed.)
Completed | 10 | 13
Not Completed | 73 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 83 | 82 | 165
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.9) | 15.5 (2.3) | 15.6 (2.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 35 | 43 | 78
  Male | 47 | 38 | 85
  Other | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 8 | 22
  Not Hispanic or Latino | 69 | 74 | 143
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 54 | 97
  Black | 26 | 20 | 46
  Asian | 1 | 1 | 2
  Mixed Race | 8 | 3 | 11
  Other | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83 | 82 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Care Inventory (SCI) Score From Baseline to 6 Months
Description: Estimate of self-management will be assessed via the Self-Care Inventory questionnaire. This scale measures self-reported adherence to diabetes self-care behaviors. A higher score on 1-5 scale is associated with more self care behaviors, i.e., better outcomes. The outcome was mean score on the scale. If a participant responded N/A, this question was not included in calculation of mean score.
Time Frame: 6 months
Population: Those analyzed were those who completed at least 1 self-care inventory survey. Analysis was preformed using multilevel mixed effects linear regression model. Outcomes are model-predicted.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 65 | 70
score on a scale | 3.57 (0.07) | 3.62 (0.07)
Statistical Analysis 1: Comparison: Intervention vs Control; A multilevel mixed effects linear regression model was used to analyze this data. This analysis allowed for an estimation of missing data. This explains the discrepancy in the number of participant study completion vs participant data analyzed (see below); Test type: Superiority — A subject was considered "completed" if they completed all 3 SCI (as indicated in participant flow section) - 13 control, 10 intervention. However, the mixed model took in to account ALL available data. As such, there were 70 control, 65 intervention that completed at least 1 SCI. Their data was analyzed by the model and used to predict later outcomes so they were considered to be included in the analysis; p = 0.035, Mixed Models Analysis — The mixed model may provide a significantly different change in SCI score from baseline to the 6 month using a per-protocol analysis in the intervention group as compared to the control group. A p value <0.05 was considered significant

2. Secondary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline to 6 Months
Description: Hemoglobin A1c is a measure of glycemic control scale that reflects how well they followed recommendations for self-care during the past month (1="never do it" to 5 ="always do this as recommended, without fail"). Total scores range from 1-70 and previous data shows that youth with better self-care levels (higher scores) have significantly better glycemic control.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-Cause Mortality and Serious Adverse Events were not monitored/assessed due to the very minimal risk of this text messaging intervention. Participants were counseled during the consent/assent process that they were eligible for the study if they had an unlimited text messaging plan, but that if that plan were to change they may begin to get charged for text messages. We asked that they reach out to us if their plan changed to avoid this event. No subjects reported this minor adverse event.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/83 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02927639/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT02927639/ICF_001.pdf